CLINICAL TRIAL: NCT04215666
Title: Diagnostic Criteria of ARDS at High Altitudes in Western China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Collaborators: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Guifen Gan, Chief physician, Affiliated Hospital of Qinghai University
Other Study IDs: ARDS Criteria high altitudes
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: ARDS
Keywords: ARDS; Definitions; high-altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild ARDS: Oxygenation standards were calculated based on the Berlin diagnostic high element correction formula combined with local atmospheric pressure
- Moderate ARDS: Oxygenation standards were calculated based on the Berlin diagnostic high element correction formula combined with local atmospheric pressure
- Severe ARDS: Oxygenation standards were calculated based on the Berlin diagnostic high element correction formula combined with local atmospheric pressure

SUMMARY:
The severity of ARDS in high altitude areas was classified according to the Berlin standard high altitude area Oxygenation.

DETAILED DESCRIPTION:
Will between January 2018 and December 2018 in lanzhou, and so on more than 1500 meters above sea level in qinghai region 10 intensive care patients with ARDS, respectively according to the standard in Berlin, Berlin, diagnosis of high altitude ARDS calibration standards and zhang the plateau region in western China put forward by the diagnosis of ALI/ARDS severity classification, observation group patients were ICU mortality, within 28 days, ICU mortality did not use breathing machine time, mechanical ventilation, ICU length of hospital stay, and the differences in hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18
* the primary disease of ARDS caused by systemic infection, shock, severe pneumonia, aspiration and trauma
* blood gas analysis showed a progressive decline in pulmonary ventilation function
* PEEP≥5cmH2O Exclusion criteria
* Receive a large amount of hormone shock therapy in a short period of time
* Died within a short time (< 24h) after mechanical ventilation
* Lack of data
* No chest imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2019 to 2022, patients diagnosed with ARDS were admitted to the department of critical care medicine of qinghai university affiliated hospital, qinghai provincial people's hospital and other selected units
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | up to 24 weeks
  mortality during treatment in ICU
28 days mortality | up to 24 weeks
  mortality at 28 days of hospitalization

SECONDARY OUTCOMES:
Ventilator Free time | up to 24 weeks
  No ventilator use time in ICU
Ventilator time | up to 24 weeks
  Ventilator time in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Gan Guifen, Bachelor, Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- Affiliated hospital of qinghai university, Xining, Qinghai, China